CLINICAL TRIAL: NCT02675465
Title: An Open-Label, Fixed-Sequence, Ascending-Dose, First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Intravenous Infusions of ATB200 Co-Administered With Oral AT2221 in Adult Subjects With Pompe Disease
Brief Title: First-In-Human Study to Evaluate Safety, Tolerability, and PK of Intravenous ATB200 Alone and When Co-Administered With Oral AT2221
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATB200-02
Record Dates: First submitted 2016-01-26; First posted 2016-02-05 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Pompe Disease
Keywords: Pompe, rhGAA
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATB200 (Experimental): Sequential single ascending doses of intravenously infused ATB200 for 3 dosing periods
  Interventions: Drug: ATB200
- ATB200 + AT2221 (Experimental): ATB200 co-administered with AT2221 (Miglustat)
  Interventions: Drug: ATB200; Drug: AT2221

INTERVENTIONS:
Drug: ATB200
  Other Names: Cipaglucosidase alfa
Drug: AT2221
  Other Names: Miglustat
  Arms: ATB200 + AT2221

SUMMARY:
This is an international, multi-center, open-label study designed to evaluate if the co-administration of investigational new drugs ATB200 and AT2221 is safe in adults with Pompe disease.

DETAILED DESCRIPTION:
This is an open-label, fixed-sequence, ascending-dose, first-in-human study to evaluate the effect of a highly targeted rhGAA (ATB200) co-administered with an enzyme stabilizer (AT2221).

The study aims to evaluate safety, tolerability, pharmacokinetics (PK), efficacy, pharmacodynamics (PD), and immunogenicity of ATB200 co-administered with AT2221.

Stage 1: evaluation of safety, tolerability, and PK following sequential single ascending doses of intravenously infused ATB200

Stage 2: evaluation of safety, tolerability, and PK following single- and multiple-ascending dose combinations of ATB200 and AT2221

Stage 3: evaluation of long term safety, tolerability, and efficacy following 24 month treatment of ATB200 co-administered with AT2221

Stage 4: open-label extension period with functional assessments every 6 months

ELIGIBILITY:
Adults with Diagnosis of Pompe disease

Cohort 1: Enzyme Replacement Therapy (ERT)-experienced subject (ambulatory):

* Male and female subjects between 18 and 65 years of age, inclusive
* Received ERT with alglucosidase alfa (Myozyme/Lumizyme) for the previous 2-6 years, inclusive
* Was receiving alglucosidase alfa at a frequency of once every other week
* Must have been able to walk 200-500 meters on the 6-Minute Walk Test (6MWT)
* Had upright Forced Vial Capacity (FVC) 30-80% of predicted normal value

Cohort 2: ERT-experienced subjects (non-ambulatory):

* Male and female subjects between 18 and 65 years of age, inclusive
* Had been receiving ERT with alglucosidase alfa for ≥2 years at a regular or set frequency
* Was wheelchair-bound

Cohort 3: ERT-naïve subjects (ambulatory):

* Male and female subjects between 18 and 65 years of age, inclusive
* Must have been able to walk 200-500 meters on the 6MWT
* Had upright FVC 30-80% of predicted normal value

Cohort 4: ERT-experienced subject (ambulatory):

* Male and female subjects between 18 and 75 years of age, inclusive
* Had been receiving ERT with alglucosidase alfa for ≥7 years, inclusive
* Was receiving alglucosidase alfa at a frequency of once every other week
* Must have been able to walk 75-600 meters on the 6MWT
* Had upright FVC 30-85% of predicted normal value

Exclusion Criteria:

* Received treatment with prohibited medications within 30 days of Baseline Visit
* Subject, if female, was pregnant or breastfeeding at screening
* Subject, whether male or female, planned to conceive a child during the study
* Had a medical or any other extenuating condition or circumstance that may, in opinion of investigator, pose an undue safety risk to the subject or compromise his/her ability to comply with protocol requirements
* Had a history of allergy or sensitivity to alglucosidase alfa, miglustat or other iminosugars (Cohorts 1, 2, and 4)
* Required invasive ventilatory support, or used noninvasive ventilatory support ≥ 6 hours a day while awake (Cohorts 1, 3, and 4)
* Had active systemic autoimmune disease such as lupus, scleroderma, or rheumatoid arthritis; subjects with autoimmune disease must have been discussed with the Amicus Medical Monitor
* Had active bronchial asthma; subjects with bronchial asthma must have been discussed with the Amicus Medical Monitor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-08-22 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (12):
  - Neuromuscular Research Centre, Phoenix, Arizona
  - University of California Irvine, Orange, California
  - University of Florida, Gainesville, Florida
  - Emory University Division of Medical Genetics, Decatur, Georgia
  - Infusion Associates, Grand Rapids, Michigan
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Abramson Cancer Center Chester County Hospital, West Chester, Pennsylvania
  - Lysosomal & Rare Disorders Research & Treatment Center (LDRTC), Fairfax, Virginia
- Womens & Childrens Hospital, Adelaide, North Adelaide, South Australia, Australia
- Germany (2):
  - University Children's Hospital Department of Neuropediatrics and Inborn Metabolic Disorders, St. Josefs-Hospital, Bochum
  - Friedrich-Baur-Institure, Dep of Neurology - University Munich, Munich
- Erasmus Medical Center, Rotterdam, Netherlands
- School of Medicine, University of Auckland, Auckland, New Zealand
- United Kingdom (2):
  - University Hospital Birmingham NHS Foundation Trust, Queen Elizabeth Medical Center, Birmingham
  - Salford Royal NHS Foundation Trust, Salford

REFERENCES:
- [Derived] Andersen H, Diaz-Manera J, Goker-Alpan O, Mozaffar T, Sitaraman Das S, Fox B, Amon F, O'Brien-Prince K, Goldman M, Holdbrook F, Jain V, Byrne BJ. Safety of home administration of cipaglucosidase alfa plus miglustat in late-onset Pompe disease: results from multiple clinical trials. Ther Adv Rare Dis. 2026 Jan 31;7:26330040261416943. doi: 10.1177/26330040261416943. eCollection 2026 Jan-Dec. PMID 41631150
- [Derived] Roberts ME, Proskorovsky I, Guyot P, Shukla P, Thibault N, Hamed A, Pulikottil-Jacob R, O'Callaghan L, Pollissard L. An Indirect Treatment Comparison of Avalglucosidase Alfa versus Cipaglucosidase Alfa Plus Miglustat in Patients with Late-Onset Pompe Disease. Adv Ther. 2025 Nov;42(11):5578-5599. doi: 10.1007/s12325-025-03301-9. Epub 2025 Sep 8. PMID 40920287
- [Derived] Byrne BJ, Schoser B, Kishnani PS, Bratkovic D, Clemens PR, Goker-Alpan O, Ming X, Roberts M, Vorgerd M, Sivakumar K, van der Ploeg AT, Goldman M, Wright J, Holdbrook F, Jain V, Benjamin ER, Johnson F, Das SS, Wasfi Y, Mozaffar T. Long-term safety and efficacy of cipaglucosidase alfa plus miglustat in individuals living with Pompe disease: an open-label phase I/II study (ATB200-02). J Neurol. 2024 Apr;271(4):1787-1801. doi: 10.1007/s00415-023-12096-0. Epub 2023 Dec 6. PMID 38057636

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 4 stages and 4 cohorts, with Stages 1 and 2 only for Cohort 1 and Stages 3 and 4 for all 4 cohorts.
Groups:
- Cohort 1 (ERT Experienced; Ambulatory): SAD 5 to 20 mg/kg ATB200: ERT experienced ambulatory subjects receiving single ascending dose (SAD) of ATB200 (5 mg/kg, 10 mg/kg, and 20 mg/kg)
- Cohort 1 (ERT Experienced; Ambulatory) MAD 20 mg/kg ATB200 + 130 to 260 mg AT2221: Enzyme replacement therapy (ERT)-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received 20 mg ATB200 in combination with 130 or 260 mg AT2221
- Cohort 1 (ERT Experienced; Ambulatory):: ERT experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received 20 mg ATB200 in combination with 260 mg AT2221
- Cohort 2 (ERT Experienced; Non-ambulatory): 20 mg/kg ATB200 + 260 mg AT2221: ERT-experienced non-ambulatory subjects with Pompe disease who had been on ERT for at least 2 years prior to enrollment. Subjects received 20 mg ATB200 in combination with 260 mg of AT2221
- Cohort 3 (ERT Naive; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221: ERT-naive ambulatory subjects with Pompe disease who were able to walk at least 200 meters in the 6MWT. Subjects received 20 mg ATB200 in combination with 260 mg of AT2221
- Cohort 4 (ERT Experienced; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for at least 7 years prior to enrollment and were able to walk at least 75 meters in the 6MWT. Subjects received 20 mg ATB200 in combination with 260 mg AT2221
Period: Stage 1 SAD (Cohort 1 Only)
Arm/Group | Cohort 1 (ERT Experienced; Ambulatory): SAD 5 to 20 mg/kg ATB200 | Cohort 1 (ERT Experienced; Ambulatory) MAD 20 mg/kg ATB200 + 130 to 260 mg AT2221 | Cohort 1 (ERT Experienced; Ambulatory): | Cohort 2 (ERT Experienced; Non-ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 3 (ERT Naive; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 4 (ERT Experienced; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221
Started | 11 | 0 | 0 | 0 | 0 | 0
Completed | 11 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2 MAD (Cohort 1 Only)
Arm/Group | Cohort 1 (ERT Experienced; Ambulatory): SAD 5 to 20 mg/kg ATB200 | Cohort 1 (ERT Experienced; Ambulatory) MAD 20 mg/kg ATB200 + 130 to 260 mg AT2221 | Cohort 1 (ERT Experienced; Ambulatory): | Cohort 2 (ERT Experienced; Non-ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 3 (ERT Naive; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 4 (ERT Experienced; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221
Started | 0 | 11 | 0 | 0 | 0 | 0
Completed | 0 | 11 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 3: 2 Year Treatment
Arm/Group | Cohort 1 (ERT Experienced; Ambulatory): SAD 5 to 20 mg/kg ATB200 | Cohort 1 (ERT Experienced; Ambulatory) MAD 20 mg/kg ATB200 + 130 to 260 mg AT2221 | Cohort 1 (ERT Experienced; Ambulatory): | Cohort 2 (ERT Experienced; Non-ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 3 (ERT Naive; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 4 (ERT Experienced; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221
Started | 0 | 0 | 11 | 6 | 6 | 6
Completed | 0 | 0 | 9 | 5 | 6 | 6
Not Completed | 0 | 0 | 2 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Stage 4: Long Term Extension
Arm/Group | Cohort 1 (ERT Experienced; Ambulatory): SAD 5 to 20 mg/kg ATB200 | Cohort 1 (ERT Experienced; Ambulatory) MAD 20 mg/kg ATB200 + 130 to 260 mg AT2221 | Cohort 1 (ERT Experienced; Ambulatory): | Cohort 2 (ERT Experienced; Non-ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 3 (ERT Naive; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221 | Cohort 4 (ERT Experienced; Ambulatory): 20 mg/kg ATB200 + 260 mg AT2221
Started | 0 | 0 | 9 | 5 | 6 | 6
Completed | 0 | 0 | 8 | 4 | 6 | 6
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6-minute walk test (6MWT)
- Cohort 2: ERT-experienced non-ambulatory subjects with Pompe disease who had been on ERT for at least 2 years prior to enrollment
- Cohort 3: ERT-naive ambulatory subjects with Pompe disease who were able to walk at least 200 meters in the 6MWT
- Cohort 4: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for at least 7 years prior to enrollment and were able to walk at least 75 meters in the 6MWT
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 11 | 6 | 6 | 6 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 5 | 5 | 26
  >=65 years | 1 | 0 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 4 | 13
  Male | 9 | 4 | 1 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 3 | 1 | 5 | 17
  Unknown or Not Reported | 3 | 3 | 5 | 1 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 3 | 1 | 5 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 5 | 1 | 12
Years since diagnosis with Pompe disease [Mean (Standard Deviation); unit: years] | 7.7 (5.11) | 15.9 (13.08) | 5.2 (4.70) | 13.0 (4.30) | 10.0 (7.98)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and Adverse Events (AEs) Leading to Discontinuation of Study Drug
Description: Number of subjects with TEAE, TESAE, and AE leading to discontinuation during the 2 year treatment period and extension (Stage 3 and 4 combined)
Time Frame: Stage 3 (2 year treatment) and Stage 4 (Extension) combined, (mean = 71 months on treatment)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg during the study.
- Cohort 2: ERT-experienced non-ambulatory subjects with Pompe disease who had been on ERT for at least 2 years prior to enrollment. Subjects received ATB200 20 mg/kg + miglustat 260 mg during the study.
- Cohort 3: ERT-naive ambulatory subjects with Pompe disease who were able to walk at least 200 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg during the study.
- Cohort 4: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for at least 7 years prior to enrollment and were able to walk at least 75 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg during the study.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 11 | 6 | 6 | 6
Participants
  Number of subjects with TEAEs | 11 | 6 | 6 | 6
  Number of subjects with TESAEs | 7 | 4 | 4 | 6
  Number of subjects with AEs leading to discontinuation | 1 | 2 | 0 | 0

2. Primary Outcome: Plasma Human Acid α-glucosidase (GAA) Activity Levels as Measured by Maximum Observed Plasma Concentration (Cmax).
Description: Plasma GAA levels (Cmax) measured in Cohorts 1 and 3 following 1st and 3rd doses of cipaglucosidase alfa + miglustat
Time Frame: 18 Weeks
Population: Pharmacokinetic (PK) analysis only performed in Cohort 1 and Cohort 3. One subject each in Cohort 1 and Cohort 3 did not have PK sample available following first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/mL/hr
Arm/Group | Cohort 1 | Cohort 3
Number analyzed (Participants) | 11 | 6
nmol/mL/hr
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st dose): number analyzed (Participants) | 10 | 5
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st dose) | 108836 (20.5) | 132400 (14.3)
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (3rd dose) | 119624 (25.7) | 105842 (15.4)

3. Primary Outcome: Plasma GAA Activity Levels as Measured by Time to Reach the Maximum Observed Plasma Concentration (Tmax).
Description: Plasma GAA levels (Tmax) measured in Cohorts 1 and 3 following 1st and 3rd doses of cipaglucosidase alfa + miglustat
Time Frame: 18 Weeks
Population: PK analysis only performed in Cohort 1 and Cohort 3. One subject each in Cohort 1 and Cohort 3 did not have PK sample available following first dose.
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 | Cohort 3
Number analyzed (Participants) | 11 | 6
h
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st Dose): number analyzed (Participants) | 10 | 5
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st Dose) | 3.49 [3.47 to 4.00] | 3.97 [3.47 to 4.00]
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (3rd Dose) | 3.57 [3.35 to 4.00] | 3.66 [3.50 to 3.98]

4. Primary Outcome: Plasma GAA Activity Levels as Measured by Area Under the Plasma Drug Concentration-time Curve (AUC).
Description: Plasma GAA levels (AUC) measured in Cohorts 1 and 3 following 1st and 3rd doses of cipaglucosidase alfa + miglustat
Time Frame: 18 Weeks
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*hr/mL
Arm/Group | Cohort 1 | Cohort 3
Number analyzed (Participants) | 11 | 6
nmol*hr/mL
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st Dose): number analyzed (Participants) | 10 | 5
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (1st Dose) | 608180 (23.7) | 762484 (22.0)
  Cipaglucosidase alfa 20 mg/kg + miglustat 260 mg (3rd Dose) | 670754 (29.4) | 638984 (18.1)

5. Secondary Outcome: Change From Baseline in 6-minute Walk Distance (6MWD)
Description: Motor function was measured in ambulatory subjects using 6MWD (meters).
Time Frame: Baseline, Month 60
Population: Motor function was evaluated using the Efficacy Population (consisting of subjects who took at least 1 dose of study drug (20 mg/kg cipaglucosidase alfa + 260 mg miglustat) and had both a baseline and at least 1 post-baseline assessment for any efficacy endpoint. 6-minute walk distance (6MWD) was only performed in ambulatory subjects (Cohorts 1, 3, and 4). Baseline and Month 60 assessment available for 9 subjects in Cohort 1, 6 subjects in Cohort 3, and 4 subjects in Cohort 4.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Cohort 1 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 9 | 6 | 4
meters | 9.2 (49.89) | -34.9 (118.80) | 27.7 (74.5)

6. Secondary Outcome: Change From Baseline in Pulmonary Function Tests
Description: Pulmonary function was measured by sitting and supine % predicted forced vital capacity (FVC)
Time Frame: Baseline, Month 60
Population: Number of participants analyzed per cohort represents the number of subjects assessed at the specific visit for the parameter. Eight subjects in Cohort 1, 1 subject in Cohort 2, and 5 subjects in Cohort 4 had FVC values reported at Month 60.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 1 | 6 | 5
percent predicted FVC
  Sitting % predicted FVC: Change from Baseline to Month 60 | -2.8 (10.93) | -8.0 (0) | 5.0 (8.07) | 3.8 (3.27)
  Supine % predicted FVC: Change from Baseline to Month 60: number analyzed (Participants) | 8 | 1 | 5 | 4
  Supine % predicted FVC: Change from Baseline to Month 60 | 0.8 (7.59) | -1.0 (0) | 1.2 (9.34) | 5.5 (5.80)

7. Secondary Outcome: Change From Baseline in Muscle Strength Tests
Description: Muscle strength was measured by total manual muscle test (MMT) score. Total MMT score ranges from 0 to 80 based on all 16 muscle groups, which are right/left shoulder abduction, right/left shoulder adduction, right/left elbow flexion, right/left elbow extension, right/left hip flexion, right/left hip abduction, right/left knee flexion, and right/left knee extension. Higher scores indicate less disease impact on muscle functions.
Time Frame: Baseline, Month 60
Population: Total MMT score was evaluated using the Efficacy Population consisting of all enrolled subjects who took at least 1 dose of study drug (20 mg/kg cipaglucosidase alfa + 260 mg miglustat co-administration) in Stage 3 and had both a baseline and at least 1 post-baseline assessment for any efficacy endpoint. Number of participants analyzed per cohort represents the number of subjects assessed at the specific visit for the parameter.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 7 | 3 | 5 | 5
score on a scale | 2.0 (5.20) | 0.0 (4.36) | 1.0 (3.54) | 3.4 (4.83)

8. Secondary Outcome: Change From Baseline in Fatigue Severity Score (FSS)
Description: The Fatigue Severity Score (FSS) consists of 9 questions, each scored on a scale from 1 ("completely disagree") to 7 ("completely agree"). The total score ranges from 9 to 63, with higher values representing higher level of fatigue due to the disease condition.
Time Frame: Baseline, Month 60
Population: The Efficacy Population consists of all enrolled subjects who took at least 1 dose of study drug (20 mg/kg cipaglucosidase alfa + 260 mg miglustat co-administration) in Stage 3 and had both a baseline and at least 1 post-baseline assessment for any efficacy endpoint. Number of participants analyzed for FSS are those in each cohort who completed the assessment at baseline and Month 60.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 3 | 6 | 4
score on a scale | 0.9 (11.48) | -4.3 (7.23) | -0.5 (8.67) | -14.0 (15.25)

9. Secondary Outcome: Change From Baseline in Overall Physical Wellbeing (Subject's Global Impression of Change [SGIC], Question1)
Description: The Subject's Global Impression of Change overall physical wellbeing (question 1) is scored on a 7-point rating scale. Improved = response of 5 or higher, No change = response of 4, and Declined = response of 3 or lower.
Time Frame: Baseline, Month 60
Population: Number of participants analyzed per cohort represents the number of subjects assessed at the specific visit for the parameter. Eight subjects in Cohort 1, 2 subjects in Cohort 2, and 5 subjects in Cohort 4 had SGIC values reported at Month 60.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 2 | 6 | 5
Participants
  Improved | 3 | 0 | 3 | 4
  No change | 2 | 2 | 1 | 0
  Declined | 3 | 0 | 2 | 1

10. Secondary Outcome: Change From Baseline in Overall Physical Wellbeing (Physician's Global Impression of Change [PGIC])
Description: The Physician's Global Impression of Change overall physical wellbeing is scored on a 7-point rating scale. Improved = response of 5 or higher, No change = response of 4, and Declined = response of 3 or lower.
Time Frame: Baseline, Month 60
Population: Number of participants analyzed per cohort represents the number of subjects assessed at the specific visit for the parameter. Eight subjects in Cohort 1, 3 subjects in Cohort 2, and 5 subjects in Cohort 4 had PGIC values reported at Month 60.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 3 | 6 | 5
Participants
  Improved | 2 | 1 | 2 | 2
  No change | 3 | 2 | 4 | 3
  Declined | 3 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected over duration of the study. Duration of participation varied by patient (range: 1.4 to 93.1 months).
Groups:
- Cohort 1: ATB200 5 mg: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received single dose of ATB200 5 mg/kg in Stage 1
- Cohort 1: ATB 200 10 mg: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received single dose of ATB200 10 mg/kg in Stage 1
- Cohort 1: ATB200 20 mg: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received single dose of ATB200 20 mg/kg in Stage 1
- Cohort 1: ATB200 20 mg + 130/260 mg Miglustat: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 130 or 260 mg in Stage 2
- Cohort 1 ATB200 20 mg/kg + Miglustat 260 mg: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for 2 to 6 years prior to enrollment and were able to walk at least 200 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg in Stage 3 and 4.
- Cohort 2 ATB200 20 mg/kg + Miglustat 260 mg: ERT-experienced non-ambulatory subjects with Pompe disease who had been on ERT for at least 2 years prior to enrollment. Subjects received ATB200 20 mg/kg + miglustat 260 mg in Stage 3 and 4.
- Cohort 3 ATB200 20 mg/kg + Miglustat 260 mg: ERT-naive ambulatory subjects with Pompe disease who were able to walk at least 200 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg in Stage 3 and 4.
- Cohort 4 ATB200 20 mg/kg + Miglustat 260 mg: ERT-experienced ambulatory subjects with Pompe disease who had been on ERT for at least 7 years prior to enrollment and were able to walk at least 75 meters in the 6MWT. Subjects received ATB200 20 mg/kg + miglustat 260 mg in Stage 3 and 4.
Arm/Group | Cohort 1: ATB200 5 mg | Cohort 1: ATB 200 10 mg | Cohort 1: ATB200 20 mg | Cohort 1: ATB200 20 mg + 130/260 mg Miglustat | Cohort 1 ATB200 20 mg/kg + Miglustat 260 mg | Cohort 2 ATB200 20 mg/kg + Miglustat 260 mg | Cohort 3 ATB200 20 mg/kg + Miglustat 260 mg | Cohort 4 ATB200 20 mg/kg + Miglustat 260 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 1/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 7/11 | 4/6 | 4/6 | 6/6
Other Adverse Events (participants affected / at risk) | 7/11 | 5/11 | 4/11 | 9/11 | 11/11 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ATB200 5 mg (N=11) | Cohort 1: ATB 200 10 mg (N=11) | Cohort 1: ATB200 20 mg (N=11) | Cohort 1: ATB200 20 mg + 130/260 mg Miglustat (N=11) | Cohort 1 ATB200 20 mg/kg + Miglustat 260 mg (N=11) | Cohort 2 ATB200 20 mg/kg + Miglustat 260 mg (N=6) | Cohort 3 ATB200 20 mg/kg + Miglustat 260 mg (N=6) | Cohort 4 ATB200 20 mg/kg + Miglustat 260 mg (N=6)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pharyngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: ATB200 5 mg (N=11) | Cohort 1: ATB 200 10 mg (N=11) | Cohort 1: ATB200 20 mg (N=11) | Cohort 1: ATB200 20 mg + 130/260 mg Miglustat (N=11) | Cohort 1 ATB200 20 mg/kg + Miglustat 260 mg (N=11) | Cohort 2 ATB200 20 mg/kg + Miglustat 260 mg (N=6) | Cohort 3 ATB200 20 mg/kg + Miglustat 260 mg (N=6) | Cohort 4 ATB200 20 mg/kg + Miglustat 260 mg (N=6)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 6 (36) | 2 (4) | 6 (43) | 4 (27)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 9 (19) | 3 (4) | 4 (5) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 1 (1) | 3 (10) | 5 (8)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (11) | 1 (1) | 4 (8) | 6 (15)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 4 (8) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (12) | 3 (3) | 4 (13) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 1 (1) | 3 (6) | 2 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 3 (5) | 5 (13)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 3 (13) | 3 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (13) | 2 (4) | 3 (8) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (23) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (1) | 3 (16) | 5 (13)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (10) | 1 (1) | 1 (1) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (11) | 0 (0) | 2 (6) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (15) | 0 (0) | 3 (5) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 1 (1) | 1 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 4 (17) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (11) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 2 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (3) | 2 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (11) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 2 (8) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 2 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 2 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (9) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (8) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (4)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (8) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Alkalosis hypochloremic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Forced vital capacity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Hypoesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza-like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Edema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilirubinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Clubbing (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Culture wound positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysstasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint noise (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoprotein (a) increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Oral viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (9) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02675465/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT02675465/SAP_001.pdf